CLINICAL TRIAL: NCT01500616
Title: Multicenter, Open-Label, Study of Telaprevir in Combination With Peginterferon Alfa and Ribavirin in Human Immunodeficiency Virus/Genotype 1 Chronic Hepatitis C Coinfected Subjects With Severe Fibrosis or Compensated Cirrhosis
Brief Title: Telaprevir Open-Label Study in Co-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018787; VX-950HPC3005 (Other: Janssen-Cilag International NV); 2011-003593-85 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic Hepatitis C Infection; Chronic Hepatitis C Co-Infected Patients; Hepatitis C; Severe Fibrosis; Compensated Cirrhosis; VX-950HPC3005
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Fibrosis | interventions — telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label telaprevir (Experimental): Depending on the patient's HAART regimen, 750 or 1125 mg telaprevir every 8 hours for 12 weeks in combination with pegylated interferon alfa and ribavirin for 48 weeks.
  Interventions: Drug: Telaprevir

INTERVENTIONS:
Drug: Telaprevir — type = exact number, unit = mg, number = 750, form = tablet, route = oral use, every 8 hours for 12 weeks in combination with pegylated interferon alfa (Peg-IFN alfa) and ribavirin (RBV) during 48 weeks for eligible non treated HIV patients and for patients whose highly active antiretroviral therapy (HAART) regimen is the combination of ritonavir-boosted atazanavir, plus either TDF or abacavir, plus either emtricitabine or lamivudine, or the combination of raltegravir, plus either TDF or abacavir, plus either emtricitabine or lamivudine, or etravirine, TDF, plus either emtricitabine or lamivudine, or etravirine, abacavir, plus either emtricitabine or lamivudine, or rilpivirine, TDF, plus either emtricitabine or lamivudine, or rilpivirine, abacavir, plus either emtricitabine or lamivudine.
Drug: Telaprevir — type = exact number, unit = mg, number = 1125, form = tablet, route = oral use, every 8 hours for 12 weeks in combination with Peg-IFN alfa and RBV during 48 weeks when patient's HAART regimen is the combination of efavirenz, plus either TDF or abacavir, plus either emtricitabine or lamivudine, or etravirine, TDF, plus either emtricitabine or lamivudine, or etravirine, abacavir, plus either emtricitabine or lamivudine, or rilpivirine, TDF, plus either emtricitabine or lamivudine, or rilpivirine, abacavir, plus either emtricitabine or lamivudine.

SUMMARY:
The purpose of this study is to collect safety and tolerability data on telaprevir treatment in combination with Peg-IFN-alfa and RBV in patients with HIV/genotype 1 chronic HCV coinfection with severe fibrosis or compensated cirrhosis who are not eligible for enrollment into an ongoing clinical study of telaprevir.

DETAILED DESCRIPTION:
In this study, all patients will receive open-label (all people involved know the identity of the intervention) telaprevir in addition to Peg IFN-alfa and RBV for treatment of hepatitis C virus (HCV) and protocol permissible treatments for HIV. Chronic hepatitis C infection causes inflammation of the liver which can potentially cause long-term complications of the current liver disease (fibrosis or cirrhosis). Therefore it is important the patient is treated for this infection. Telaprevir is an experimental medication that has been tested for the treatment of hepatitis C infections in several previous studies in more than 2500 patients. Telaprevir is a member of a new class of drugs being developed for chronic hepatitis C: Direct Acting Antiviral (DAA) agents. Unlike pegylated interferon (Peg-IFN) and ribavirin (RBV), DAA agents act directly on the hepatitis C virus (HCV) replication cycle. The aim of the telaprevir treatment is to eradicate the Hepatitis C virus out of the patient's body. This can be measured by testing the amount of a certain part of this Hepatitis C virus, called the Ribonucleic acid (RNA [HCV RNA]) in their blood. It is possible that the patient will not respond to the therapy and the levels of HCV RNA in their blood will not decrease or even increase. Based on these results it might be decided the patient will not benefit from treatment and he/she need to stop the telaprevir only or all medication for their hepatitis C infection. The doctor will keep them informed about the patient's reaction to the treatment and will take the necessary measurements as prescribed by the study protocol and routine medical practice. During the study the patient will simultaneously be treated with the therapy that the doctor would normally prescribe for treatment of their chronic hepatitis C infection: "ribavirin (RBV)" and "pegylated interferon alfa (PEG-INF-alfa)". Telaprevir is always administered in combination with RBV and PEG-IFN-alfa. In function of the patient's specific HIV status, the doctor has prescribed, or not, a specific treatment that the patient will continue to take during the study. This treatment could be: (a) efavirenz, tenofovir disoproxil fumarate (TDF), plus either emtricitabine or lamivudine, (b) efavirenz, abacavir, plus either emtricitabine or lamivudine, (c) ritonavir-boosted atazanavir, TDF, plus either emtricitabine or lamivudine, (d) ritonavir-boosted atazanavir, abacavir, plus either emtricitabine or lamivudine, (e) raltegravir, TDF, plus either emtricitabine or lamivudine, (f) raltegravir, abacavir, plus either emtricitabine or lamivudine or (g) etravirine, TDF, plus either emtricitabine or lamivudin, (h) etravirine, abacavir, plus either emtricitabine or lamivudine, (i) rilpivirine, TDF, plus either emtricitabine or lamivudine, (j) rilpivirine, abacavir, plus either emtricitabine or lamivudine, (k) no treatment. In an interim analysis of a Phase 2a study, human immunodeficiency virus (HIV)-1/HCV genotype 1 coinfected patients currently receiving HIV therapy who had telaprevir added to Peg IFN-alfa-2a and RBV regimen for treatment of their HCV genotype 1 infection had a higher HCV RNA response (undetectable HCV RNA) at Weeks 4 and 12 than those who received only the Peg-IFN-alfa-2a and RBV regimen. These responses were sustained through Week 24, with 73.7% of patients who had telaprevir added to the Peg-IFN-alfa-2a and RBV regimen and 54.5% of patients who received only the Peg-IFN-alfa-2a and RBV regimen also achieving undetectable HCV RNA at Week 24. Patients with severe fibrosis or cirrhosis have a lower likelihood of sustained virologic response (SVR) and also have the greatest risk of liver failure, hepatocellular carcinoma (HCC), and death. Administering telaprevir in this difficult to treat population may reduce the risk of long-term complications associated with HCV in patients with HIV/HCV genotype 1 coinfection. All patients eligible to enter the study will receive telaprevir (750 or 1,125 mg every 8 hours based on their Highly Active Antiretroviral Therapy (HAART) regimen) during the first 12 weeks of the study in combination with Peg IFN alfa/RBV. Patients will subsequently be treated with Peg-IFN-alfa/RBV for an additional 36 weeks. The total duration of Peg-IFN-alfa/RBV will be 48 weeks. HCV RNA levels should be measured at Weeks 4, 12, 24 and 48. All patients should have a posttreatment follow-up visit, including measurement of plasma HCV RNA levels, performed 24 weeks after the last administered dose of treatment. Note that in certain countries, an additional main objective of the study is to provide Early Access to telaprevir in this population.

ELIGIBILITY:
Inclusion Criteria: - Have diagnosis of HIV-1 or HIV-2 infection, or HIV-1 and HIV-2 coinfection for more than 6 months before the screening visit. - Should have been on a stable permissible HAART regimen for more than 8 weeks before Day 1 without switches. OR Not on a HAART regimen and not expected to start HIV treatment during the study, ie, have CD4 count of ≥500 cells/mm3 and a HIV-1 and/or HIV-2 viral load ≤50,000 copies/mL at screening - If on stable permissible HAART regimen, have CD4 count ≥200 cells/mm3 or ≥15% and HIV-1 and/or HIV-2 viral load <50 copies/mL for at least 6 months before starting treatment is recommended - Have evidence of HCV infection genotype 1 (molecular assay) - Have a quantifiable plasma HCV RNA Exclusion Criteria: - Is eligible for enrollment into an ongoing clinical study of telaprevir - Is infected or coinfected with HCV of another genotype than genotype 1 - Has a contraindication to the administration of Peg-IFN-alfa or RBV, or medical history or laboratory values that preclude treatment with Peg-IFN-alfa or RBV according to the respective local prescribing information - Have any contraindication to the currently prescribed HAART regimen at screening. Note: Patients who have a contraindication to a nonprescribed permissible HAART medication are not excluded. - Positive human leukocyte antigen (HLA)-B5701 genotyping result at screening (or documented result prior to screening) if abacavir is a component of HAART

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events | from first use of the medicinal product to 30 days after administration of the last dose of investigational product (telaprevir)
  Protocol-defined adverse events whether serious or non-serious, that occur from the first use of investigational product (telaprevir) to 30 days after administration of the last dose of investigational product (telaprevir) will be part of the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV, Belgium Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (29):
- Belgium (6):
  - Antwerp
  - Brussels
  - Charleroi
  - Ghent
  - Leuven
  - Liège
- Germany (8):
  - Berlin
  - Bonn
  - Cologne
  - Dortmund
  - Frankfurt
  - Hanover
  - Stuttgart
  - Tübingen
- Budapest, Hungary
- Dublin, Ireland
- Luxembourg, Luxembourg
- Portugal (3):
  - Amadora
  - Lisbon
  - Porto
- Russia (5):
  - Perm
  - Saint Petersburg
  - Tolyatti
  - Volgograd
  - Yoshkar-Ola
- United Kingdom (4):
  - Glasgow
  - Liverpool
  - London
  - Plymouth

REFERENCES:
- [Derived] Gori A, Doroana M, Chernova O, Rockstroh JK, Banhegyi D, Bergin C, Verucchi G, Liu C, DeMasi R, Hadacek B, Nelson M. Telaprevir-based therapy for treatment of HIV-1 and hepatitis C virus co-infected patients: An early access programme. J Infect. 2015 Dec;71(6):675-82. doi: 10.1016/j.jinf.2015.09.013. Epub 2015 Sep 28. PMID 26416471
- See also: Multicenter, Open-Label Study of Telaprevir in Combination With Peginterferon Alfa and Ribavirin in Human Immunodeficiency Virus/Genotype 1 Chronic Hepatitis C Coinfected Subjects With Severe Fibrosis or Compensated Cirrhosis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3335&filename=CR018787_CSR.docx